CLINICAL TRIAL: NCT02407665
Title: A Pilot fMRI Study of Fibromyalgia: Tai Chi Intervention
Brief Title: Tai Chi Intervention and Brain Imaging Study Among Fibromyalgia Patients and Healthy Controls
Acronym: fMRI/FMEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11552
Record Dates: First submitted 2015-03-18; First posted 2015-04-03 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Fibromyalgia; Chronic Pain
Keywords: Tai Chi; fMRI
MeSH Terms: conditions — Fibromyalgia; Chronic Pain | interventions — Tai Ji

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tai Chi (Experimental): Participants who practice Tai Chi 2X/week for 12-weeks
  Interventions: Behavioral: Tai Chi
- Healthy Control (No Intervention): 24 healthy controls

INTERVENTIONS:
Behavioral: Tai Chi — Each Tai Chi session will last 60 minutes and will continue twice a week for 12 weeks. Our instructors, who have extensive experience conducting Tai Chi training programs, will follow the standardized Tai Chi protocol. We will also provide the participants with printed materials on FM and the Tai Chi Mind-Body program, including Tai Chi principles, practicing techniques, and safety precautions for participants with FM
  Arms: Tai Chi

SUMMARY:
This exploratory study proposal is the first pilot brain imaging study to determine if Tai Chi can modulate brain resting state functional connectivity (rsFC) and brain morphometry among fibromyalgia (FM) patients and healthy controls.

DETAILED DESCRIPTION:
Twenty-four FM patients and 24 age matched healthy control will be recruited. All FM patients will undergo Tai Chi intervention twice weekly for 12 weeks of practice. fMRI resting state and brain structure data will be collected before and after treatment. For the healthy control group, the fMRI and structure data will only be collected once, contemporaneous with the 12 week scan for the fibromyalgia patients.

The primary outcome will be rsFC of rostral anterior cingulate cortex (rACC), a key region in descending pain modulatory system (DPMS). The secondary outcome include change of the cortical thickness changes, fibromyalgia symptom severity, widespread pain index, depression, stress/anxiety, sleep quality, and quality of life. Covariates include age, gender, body mass index, disease duration, depression, and comorbidities. Clinical outcome measurements will be collected at baseline and after 12 weeks of intervention for the fibromyalgia cohort and at a single visit for the healthy controls. The Tai Chi classes will be taught at Tufts Medical Center and the fMRI scans will be performed at Massachusetts General Hospital Martinos Center.

The project will advance science in the field of mind-body medicine for chronic pain management, both mechanistically and clinically.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years or older.
* Fulfills the American College of Rheumatology (ACR) 1990 classification criteria for FM: (1) a history of widespread musculoskeletal pain on the right and left sides of the body as well as above and below the waist for a minimum duration of 3 months, and (2) pain in 11 or more of 18 specific tender points with moderate or greater tenderness reported upon digital palpation.22
* Fulfills the ACR 2010 diagnostic criteria for FM: (WPI ≥7 AND SS ≥5) OR (WPI 3-6 AND SS ≥9) and does not have a disorder that would otherwise explain the pain23
* Willing to complete a 12-week, twice-a-week Tai Chi exercise program.
* Willing to abstain from Aerobic Exercise or other new formalized exercise programs until completion of the study.
* Willing to undergo MRI at baseline and follow-up.

Exclusion Criteria:

* Prior experience with Tai Chi or other similar types of Complementary and Alternative Medicine in the past 1 year such as Qi gong and yoga since these share some of the principles of Tai Chi.
* Dementia, neurological disease, cancer, cardiovascular disease, pulmonary disease, metabolic disease, renal disease, liver disease, or other serious medical conditions limiting ability to participate in the Tai Chi programs, as determined by the study physicians.
* Any other diagnosed medical condition known to contribute to FM symptomatology, such as thyroid disease, inflammatory arthritis, systemic lupus erythematosis, rheumatoid arthritis, myositis, vasculitis or Sjogren's syndrome.
* Inability to pass the Physical Activity Readiness Questionnaire (PAR-Q)
* Inability to pass the Mini-Mental Status examination (with a score below 24)24 Enrollment in any other clinical trial within the last 30 days
* Plan to permanently relocate from the region during the trial period
* Presence of any contraindications to fMRI scanning. Including but not limited to: cardiac pacemaker, metal implants, fear of closed spaces, pregnancy, weight >300 lbs
* Non-English Speaking.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Brain Resting State Functional Connectivity as measured by fMRI | Modulation of impaired rsFC and brain structure at 12 weeks
  rostral anterior cingulate cortex (rACC), a key region in descending pain modulatory system (DPMS)

SECONDARY OUTCOMES:
Cortical Thickness as measured by fMRI | Baseline and 12-week
Fibromyalgia Symptom Severity as measured by FIQR Questionnaire | Baseline, weekly, and 12-week
  FIQR
Widespread Pain Index as measured by Clinical Diagnostic Criteria for Fibromyalgia Questionnaire | Baseline and 12-week
  Clinical Diagnostic Criteria for Fibromyalgia
Depression as measured by BECK-II Questionnaire | Baseline and 12-week
  BECK-II
Stress/Anxiety as measured by Hospital Anxiety and Depression Scale | Baseline and 12-week
  Hospital Anxiety and Depression Scale
Sleep Quality as measured by PSQI Questionnaire | baseline and 12-week
  PSQI
Quality of Life as measured by visual analog scale and SF-36 Questionnaire | baseline and 12-week
  VAS, SF-36
Mindfulness as measured by Five Facet Mindfulness Questionnaire | baseline and 12-week
  FFMQ
Self-Efficacy as by Chronic Pain and Self Efficacy Questionnaire | baseline and 12-week
  Chronic Pain Self Efficacy
Quantitative Sensory Testing as measured by an Algometer | baseline and 12-week
  Pain threshold

CONTACTS AND LOCATIONS:
Overall Officials: Chenchen Wang, MD, MSc, Principal Investigator — Tufts University School of Medicine
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kong J, Huang Y, Liu J, Yu S, Ming C, Chen H, Wilson G, Harvey WF, Li W, Wang C. Altered functional connectivity between hypothalamus and limbic system in fibromyalgia. Mol Brain. 2021 Jan 20;14(1):17. doi: 10.1186/s13041-020-00705-2. PMID 33472674